CLINICAL TRIAL: NCT02123316
Title: Assessment of the Effectiveness of a Dermatophagoides Pteronyssinus Extract, Rated in Units of Mass and Administered Subcutaneously for the Treatment of Local Allergic Rhinitis. Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Subcutaneous Immunotherapy With Dermatophagoides Pteronyssinus in Local Allergic Rhinitis
Acronym: ECRL1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Miguel Blanca Gomez (Other)
Responsible Party: Sponsor-Investigator, Miguel Blanca Gomez, MD, Plaza del Hospital Civil
Organization: Plaza del Hospital Civil (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECRL12008-003680-39; 2008-003680-39 (EudraCT Number)
Record Dates: First submitted 2014-04-19; First posted 2014-04-25 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2014-04

CONDITIONS: Local Allergic Rhinitis
Keywords: local allergic rhinitis; subcutaneous immunotherapy; house dust mite allergy; Dermatophagoides pteronyssinus allergy
MeSH Terms: conditions — Dust Mite Allergy | interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pangramin Plus D. pteronyssinus (Active Comparator): Pangramin Plus D. pteronyssinus 100% for subcutaneous injection
  Interventions: Biological: Pangramin Plus D. pteronyssinus
- Placebo (Placebo Comparator): Placebo for subcutaneous injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Pangramin Plus D. pteronyssinus — Subcutaneous immunotherapy with Dermatophagoides pteronyssinus
  Arms: Pangramin Plus D. pteronyssinus
Biological: Placebo — Placebo for subcutaneous injection
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of an extract of Dermatophagoides pteronyssinus versus placebo in the treatment of local allergic rhinitis. The primary efficacy endpoint is the reduction in symptom scores and medication use in the active group compared to placebo.

The influence of treatment in "in vitro" and "in vivo" objective parameters was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Prior to study specific examinations the patient has to give his/her written informed consent.
* Local allergic rhinitis induced by Dermatophagoides pteronyssinus (DP).
* Age: 18-55.
* Negative skin prick-test to DP
* Positive nasal allergen provocation test to DP (NAPT-DP) and/or nasal specific IgE (sIgE) to DP>0.35 kU/L
* If applicable negative urine pregnancy test and willingness to use effective form of contraception for the duration of involvement in the study.

Exclusion Criteria:

* Severe immunopathological or immunodeficiencies diseases.
* Treatment with beta-blockers, even when administered topically
* Severe psychological disorders
* Severe Atopic Dermatitis
* FEV1 <70% predicted after appropriate pharmacological treatment
* History of hypersensitivity or intolerance to excipients and / or trial medication or other medication to be used for protocol
* Inability to adequately perform diagnostic tests or treatment
* Awareness of other inhaled allergens (perennial or seasonal) clinically relevant to the subject and that may interfere with the response evaluation
* Treatment with immunotherapy in the 5 years prior to his inclusion in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Symptoms-Medication score at 1,3,6,12,18, and 24 months | Baseline, month 1,3,6,12,18, and 24
  Patients were provided a diary to score the severity of their symptoms and the use of rescue medication during 4 consecutive weeks.
  Nasal symptoms of rhinorrhea, nasal congestion, sneezing, nasal itching, and ocular symptoms were recorded using a 4-point categorical scale from 0 to 3 (0: no symptoms, 1:mild, 2:moderate; 3:severe).
  The use of rescue medication was recorded in the patient diary according to the following score:
  Oral antihistamines (1 tablet = 1 point); intranasal corticosteroids (400mcg/day of beclometasone or equivalent = 1.4 points); and ocular antihistamines (1 dose = 1 point).

SECONDARY OUTCOMES:
Change from Baseline response skin prick-test at 1,3,6,12,18, and 24 months | Baseline, month 1,3,6,12,18, and 24
Change from Baseline response to intradermal test at 1,3,6,12 and 24 months | Baseline, month 1,3,6,12,18, and 24
Change from Baseline flow cytometry study at 1,3,6,12,18, and 24 months | Baseline, month 1,3,6,12,18, and 24
Change from Baseline determination of tryptase, eosinophilic cationic protein, IgG, IgG4 and specific D. pteronyssinus-IgE by Immunoassay at 1,3,6,12,18, and 24 months | Baseline, month 1,3,6,12,18 and 24
Change from Baseline response to nasal allergen provocation test with Dermatophagoides pteronyssinus at 1,3,6,12,18 and 24 months | Baseline, month 1,3,6,12,18 and 24
Adverse event | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Blanca, MD, PhD, Principal Investigator — Allergy Unit, Regional University Hospital of Malaga, Spain
Locations (1):
- Hospital Carlos Haya, Málaga, Malaga, Spain

REFERENCES:
- [Derived] Rondon C, Campo P, Salas M, Aranda A, Molina A, Gonzalez M, Galindo L, Mayorga C, Torres MJ, Blanca M. Efficacy and safety of D. pteronyssinus immunotherapy in local allergic rhinitis: a double-blind placebo-controlled clinical trial. Allergy. 2016 Jul;71(7):1057-61. doi: 10.1111/all.12889. Epub 2016 Apr 13. PMID 27008542